CLINICAL TRIAL: NCT03711708
Title: A PHASE IV, SINGLE-DOSE, OPEN-LABEL, RANDOMIZED, 2-WAY CROSSOVER STUDY TO DETERMINE THE RELATIVE BIOAVAILABILITY OF ZOLOFT (REGISTERED) ORAL SOLUTION (20 MG/ML; FARMASIERRA MANUFACTURING, S.L.) COMPARED TO ZOLOFT (REGISTERED) TABLETS (50 MG; WYETH INDÚSTRIA FARMACÊUTICA LTDA.) IN HEALTHY RESEARCH SUBJECTS UNDER FASTED CONDITIONS
Brief Title: Relative Bioavailability Study of Zoloft Oral Solution to Zoloft Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0501107
Record Dates: First submitted 2018-10-01; First posted 2018-10-18 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zoloft Oral Solution (Experimental): 50 mg sertraline administered as 2.5 mL of Zoloft Oral Solution (20 mg/mL) after dilution with 120 mL of water.
  Interventions: Drug: Zoloft Oral Solution
- Zoloft Tablets (Active Comparator): Zoloft 50 mg tablet.
  Interventions: Drug: Zoloft tablets

INTERVENTIONS:
Drug: Zoloft Oral Solution — Test Product: 50 mg sertraline administered as 2.5 mL of Zoloft Oral Solution (20 mg/mL) after dilution with 120 mL of water
  Arms: Zoloft Oral Solution
Drug: Zoloft tablets — Reference Product: 50 mg sertraline administered as 1x Zoloft 50 mg tablet
  Arms: Zoloft Tablets

SUMMARY:
In Brazil, sertraline is currently available as film coated tablets for oral administration containing sertraline hydrochloride equivalent to 50 mg or 100 mg sertraline.

The sponsor has developed an oral solution formulation containing 20 mg/mL of sertraline, which must be diluted with 120 mL of water, ginger ale, lime/lemon soda or orange juice to be palatable before use. The purpose of this study is to evaluate the relative bioavailability of Zoloft oral solution compared to Zoloft tablets in healthy participants under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female research subjects and/or male research subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.
* Female research subjects of non-childbearing potential
* Body mass index (BMI) of 18.5 kg/m2 to 24.9 kg/m2, and a total body weight >50 kg (>110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the research subject has been informed of all pertinent aspects of the study.
* Research subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Clinically significant infections within the past 3 months, evidence of any infection within the past 7 days, history of disseminated herpes simplex infection or recurrent (>1 episode) or disseminated herpes zoster.
* Evidence or history of cyclic neutropenia.
* Personal or family history of hereditary immunodeficiency (eg, severe combined immunodeficiency disorder [SCID], Wiskott Aldrich syndrome, X linked agammaglobulinemia).
* Vaccination with live or attenuated vaccines within 6 weeks prior to dosing, or is to be vaccinated with these vaccines at any time during treatment or within 6 weeks following discontinuation of dosing.
* Any condition possibly affecting drug absorption (eg, gastrectomy, colon resection, etc.).
* Research subjects with a history of, or current evidence for, severe gastrointestinal narrowing (pathologic or iatrogenic).
* History of or current positive results for any of the following serological tests: hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), anti hepatitis C core antibody (HCV Ab), or human immunodeficiency virus (HIV) 1 and 2.
* A positive urine drug test.
* A positive alcohol screen.
* History of regular alcohol consumption exceeding 14 drinks/week for female research subjects or 21 drinks/week for male research subjects [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months before screening.
* Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day. For chewing tobacco, one chew is equivalent to approximately 2 3 cigarettes, so research subjects would be limited to 2 or less chews per day.
* Treatment with an investigational drug within 6 months or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Pregnant female research subjects, breastfeeding female research subjects, fertile male research subjects and female research subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol from at least 14 days prior to the first dose of investigational product until at least 28 days after the last dose of investigational product.
* A positive beta human chorionic gonadotropin test for women of childbearing potential.
* Use of prescription or nonprescription drugs and dietary supplements within 14 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.
* Herbal supplements, hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone releasing intrauterine devices [IUDs], vaginal ring, and postcoital contraceptive methods), and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product.
* Depo Provera must have been discontinued at least 6 months prior to the first dose of investigational product.
* Consumption of grapefruit or grapefruit related citrus fruits (eg, Seville oranges, pomelos) or juices within 7 days prior to dosing.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 3 months prior to screening.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* History of hypersensitivity to sertraline or any of the components in the formulation of the study products.
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the research subject inappropriate for entry into this study.
* Research subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or research subjects who are the sponsor's employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Area under the sertraline plasma concentration-time curve from time zero to last time point (AUClast) | Predose (0 h), at 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 10, 12, 24, 48, 72, 96, 120, and 144 hours post dose
Maximum observed plasma concentration of sertraline (Cmax) | Predose (0 h), at 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 10, 12, 24, 48, 72, 96, 120, and 144 hours post dose

SECONDARY OUTCOMES:
Time to first occurrence of Cmax (Tmax) of sertraline | Predose (0 h), at 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 10, 12, 24, 48, 72, 96, 120, and 144 hours post dose
Sertraline plasma elimination half life (t½) | Predose (0 h), at 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 10, 12, 24, 48, 72, 96, 120, and 144 hours post dose
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 144 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICF - Instituto de Ciencias Farmaceuticas de Estudos e Pesquisas Ltda, Aparecida de Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501107&StudyName=A+Phase+Iv%2C+Single-dose%2C+Open-label%2C+Randomized%2C+2-way+Crossover+Study+To+Determine+The+Relative+Bioavailability+Of+Zoloft+%28registered%29+Oral+Solution+%2820+Mg%2Fml%3B+Farmasierra+Manufacturing%2C+S.l.%29+Compared+To+Zoloft+%28registered%29+Tablets+%2850+Mg%3B+Wyeth+Ind%C3%BAstria+Farmac%C3%AAutica+Ltda.%29+In+Healthy+Research+Subjects+Under+Fasted+Conditions
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501107&StudyName=A+PHASE+IV%2C+SINGLE-DOSE%2C+OPEN-LABEL%2C+RANDOMIZED%2C+2-WAY+CROSSOVER+STUDY+TO+DETERMINE+THE+RELATIVE+BIOAVAILABILITY+OF+ZOLOFT+%28REGISTERED%29+ORAL+SOLUTION+%2820+MG%2FML%3B+FARMASIERRA+MANUFACTURING%2C+S.L.%29+COMPARED+TO+ZOLOFT+%28REGISTERED%29+TABLETS+%2850+MG%3B+WYETH+IND%C3%9ASTRIA+FARMAC%C3%8AUTICA+LTDA.%29+IN+HEALTHY+RESEARCH+SUBJECTS+UNDER+FASTED+CONDITIONS